CLINICAL TRIAL: NCT02701829
Title: Taxi METERS: Measuring Effectiveness of Technology, Education, Referrals and Support
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 16-038
Record Dates: First submitted 2016-03-02; First posted 2016-03-08 (Estimated); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Improving Blood Pressure Control
Keywords: taxi cab drivers; high blood pressure; 16-038
MeSH Terms: conditions — Hypertension | interventions — Health Fairs; PLEKHG5 protein, human

ARMS (3):
- Health Fairs (HF) (Experimental): Drivers will undergo U&C Health Fair follow-up either Regular or Urgent Follow-up: Timeline is determined by health status, with regular follow-up continuing for at least two weeks and urgent follow-up continuing for at least a month
  Interventions: Other: CONTROL- Usual & Customary Health Fair Follow-up
- HF + text messaging + home BP monitoring (Experimental): Drivers will receive: U&C HF follow-up, Mobile text messaging intervention w/ interactive 2- way messaging to encourage BP management for nine months A home BP monitoring equipment with instructions to self-monitor BP for nine months
  Interventions: Other: Health Fair + TECH [Text Messaging + Home Blood Pressure Monitoring]
- HF +Tech + social network support (SNS). (Experimental): Drivers will receive:
  U&C HF follow-up, Mobile text messaging intervention w/ interactive 2- way messaging to encourage BP management for nine months and home BP monitoring equipment with instructions to self-monitor BP for nine months A social network support intervention in which selected family/peers encourage drivers to maintain healthy behaviors for nine months
  Interventions: Other: Heal th Fair + TECH [Text Messaging + Home Blood Pressure Monitoring] + Social Network Support (SNS)

INTERVENTIONS:
Other: CONTROL- Usual & Customary Health Fair Follow-up — participating drivers may fall into 1 of 2 categories- Regular follow-up, or Urgent Follow-up.
  Arms: Health Fairs (HF)
Other: Health Fair + TECH [Text Messaging + Home Blood Pressure Monitoring] — all participating drivers receives standard Health Fair services initially falling into 1 of 2 categories-Regular Follow-up or Urgent Follow-up. Additionally all participating drivers will receive Home Blood Pressure Monitors and have the mobile health text messaging intervention.
  Arms: HF + text messaging + home BP monitoring
Other: Heal th Fair + TECH [Text Messaging + Home Blood Pressure Monitoring] + Social Network Support (SNS) — all participating drivers receives standard Health Fair services initially falling into 1 of 2 categories-Regular Follow-up or Urgent Follow-up. Additionally all participating drivers will receive Home Blood Pressure Monitors for daily BP self-monitoring and text messaging, and they will receive the social network support intervention including an SNS guide for each SNS.
  Arms: HF +Tech + social network support (SNS).

SUMMARY:
In our past work it was found that many drivers had high blood pressure, and lifestyles that led to being overweight and not having cancer screenings performed. The investigators are now adding to the Health Fairs' usual program different ways of following up with drivers who attend our Health Fairs. The investigators are doing this because they want to find the best way to help drivers manage high blood pressure, and reduce cancer risk, by maintaining a healthy weight and increasing colorectal cancer screening. Health screenings will be conducted by trained personnel, and a physician or nurse will provide a health consult in person or over the phone (via MSK-issued phone/video/audio devices).

In the event that participants are unable to meet in person for biometric measurements, staff will accept their self-reported weight, blood pressure, and waist circumference over the phone. Staff may mail blood pressure machines (to participants who did not receive them at baseline), scales, and measuring tapes to participants to assist in the completion of self-reported biometric measures. Along with supplies, participants may also receive a letter asking for the confirmation of supply receipt.

* If critically abnormal values are identified during the health fair, under the advisement of the clinician, the driver may be escorted by trained staff directly to a health care facility for immediate medical follow-up

ELIGIBILITY:
Inclusion Criteria:

* Male
* Hypertensive-level readings over three weeks, with at least two of three elevated BP readings (systolic ≥140 and/or diastolic ≥90); OR
* One hypertensive crisis readings (systolic ≥165 and/or diastolic ≥100) {eligible for the study without having to return for second or third readings} OR
* have a known diagnosis of hypertension and have elevated values at one reading {eligible for the study without having to return for second or third readings}
* Over 19 years of age (we are selecting participants older than three years past the legal driving age of 16, as younger drivers tend to change jobs more often);
* Planning on remaining in NYC for at least 9 months (with no vacations or trips to exceed two months)
* Licensed taxi driver for at least 3 months;
* Speaks English, Spanish, Bengali, Urdu, or French;
* Owns a cell phone that can receive text messages and is willing to receive text messages for this study

Exclusion Criteria:

* Part-time driver (drives fewer than 35 hours per week). Although it is highly unlikely for NYC taxi drivers to work for multiple garages at study baseline, drivers may switch jobs and/or their garage base affiliation while participating in this study. New jobs and/or garage base affiliations will be tracked during follow-up assessments and noted for potential limitations with study retention and intervention contamination. Drivers will be allowed to continue the study even if they are no longer working with the initial garage base.
* Driver currently has (or has a history of) any CVD including coronary artery disease, angina or aortic stenosis; this does not include hypertension.

Min Age: 21 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2025-10-27 (Actual); Study Completion 2025-10-27 (Actual)

PRIMARY OUTCOMES:
decrease in blood pressure levels | 9 months
  The drop in BP from baseline will be estimated for each participant. The investigators will summarize the mean and 95% confidence interval (CI) for the drop in systolic and diastolic BP from baseline for each arm at the

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Gany, MD, MS, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/